CLINICAL TRIAL: NCT00605592
Title: UVA Islet Cell Transplantation in Patients With Type I Diabetes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Kenneth Brayman/MD, PhD, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12839
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 Diabetes; Kidney Transplant; Hypoglycemic Unawareness; Islet Transplant; Pancreatic Islet Cell Transplantation; University of Virginia; Islet Transplantation; Kidney Transplantation
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Islet cell transplant
  Interventions: Procedure: Pancreatic Islets of Langerhans Cell Transplant

INTERVENTIONS:
Procedure: Pancreatic Islets of Langerhans Cell Transplant — Transplantation of islet cells will be given to eligible patients, up to three times during the study, using cell quantities based on body weight.
  Other Names: Islet Cell Transplant; Pancreatic Islet Cell Transplantation

SUMMARY:
This protocol will provide islet cell transplantation to two separate populations in need of a pancreas transplant:

Group I: Islet Cell Transplantation in Type I Diabetics without Kidney Problems

Group II: Islet Cell Transplantation in Type I Diabetics Who Have a Stable Functioning Kidney Transplant

The targeted patients have very brittle diabetes or dangerous hypoglycemic unawareness and may benefit from transplantation over continuing insulin therapy, even though chronic immunosuppression is required. We believe that in these patients, the islet transplant procedure promises enough potential benefit to justify subjecting patients who have not previously had a transplant to the risk of immunosuppression.

In patients who are already subject to the dangers of chronic immunosuppression for other reasons, i.e. to prevent rejection of a kidney allograft, the islet transplantation procedure itself is the principal additional risk and this risk should be minimal. In these patients (our Group II), the potential benefit from improved glycemic control is that it promises to slow or even reverse diabetic complications, such as vascular problems leading to kidney damage. It is this rationale that has made pancreas transplantation a widely accepted option in patients with renal failure, despite the risks associated with whole pancreas transplantation. Islet cell transplantation aims to provide a potentially lower risk procedure that has similar relief from diabetic complications.

ELIGIBILITY:
Inclusion Criteria:

* Type I Diabetes Mellitus for at least 5 years
* Unstable control of diabetes despite intensive care by an endocrinologist, including episodes of dangerously low blood sugars
* Group I must have healthy kidneys
* Group II (islet after kidney) must have a stable kidney allograft for at least 6 months

Exclusion Criteria:

* Unstable diabetic eye disease
* Poor kidney function
* Type II Diabetes as determined by blood tests
* Any history of cancer, except certain skin cancers
* Pregnant or unwilling to use adequate birth control
* Very high hemoglobin A1c levels
* Poor control of blood pressure, despite use of medications
* Very high insulin requirements
* History of exposure to HIV
* Active Hepatitis B or Hepatitis C infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
A decrease in the average daily insulin requirement post-islet cell transplantation. | Post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Brayman, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States